CLINICAL TRIAL: NCT02126254
Title: Optimization of the Treatment of Acute Heart Failure by a Non Invasive Cardiac System-Randomized Control Trial
Brief Title: Optimization of the Treatment of Acute HF by a Non Invasive Cardiac System-a Randomized Control Trial
Acronym: HFNICAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, michal roll, Tel-Aviv Medical Center, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-14-YA-055-CTIL
Record Dates: First submitted 2014-04-22; First posted 2014-04-29 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Heart Failure; Kidney Injury
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Control group will be treated in the cardiology and internal medicine departments according to the guidelines for the management of Heart Failure
- Hemodynamic group (Active Comparator): Hemodynamic group patients will be examined in the cardiology and internal medicine departments and treated according to the NICaS system in addition to current guidelines. Patients in this group will be tested within 12 hours from hospitalization and thereafter on an everyday basis until discharge
  Interventions: Device: Hemodynamic group

INTERVENTIONS:
Device: Hemodynamic group — NICAS guided treatment
  Arms: Hemodynamic group

SUMMARY:
The aim of this trial is to compare the efficacy of NICaS-directed treatment strategy to the common treatment strategy (based on clinical judgment) on morbidity and mortality in patients with decompensated congestive heart failure, and accordingly to assess whether the NICaS system can optimize and individualize the treatment of decompensated heart failure patients. A prospective randomized controlled trial in which Known HF patients, with reduced EF <40%, admitted due to decompensated HF, will be randomly assigned, in a 1:1: ratio, to either: 1) Control group that will be treated in the cardiology and internal medicine departments according to the guidelines for the management of Heart Failure. 2) Hemodynamic group patients will be examined in the cardiology and internal medicine departments and treated according to the NICaS system in addition to current guidelines. Patients in this group will be tested within 12 hours from hospitalization and thereafter on an everyday basis until discharge. For all patients randomized, therapy will be tailored to the ultimate goal of discharge on an oral medical regimen to provide better relief of CHF symptoms, to reduce filling pressures and to maintain adequate perfusion. These goals are the same for both groups, but in the control group therapy will be adjusted according to clinical assessment alone, while in the NICaS-directed group, actual measurement of hemodynamics will be used to supplement clinical assessment.

DETAILED DESCRIPTION:
Heart failure is a complex clinical syndrome that results from any structural or functional impairment of ventricular filling or ejection of blood. Although survival has improved, the absolute mortality rates for HF remain approximately 50% within 5 years of diagnosis. In the ARIC study, the 30-day, 1-year, and 5-year mortallity rates after hospitalization for HF were 10.4%, 22%, and 42.3%, respectively. HF represents a major burden in the developed world. In the United States, HF is the primary diagnosis for more than 1 million hospitalized patients annually. A significant number of patients with acute decompensated heart failure have baseline renal insufficiency. Yet perhaps more important is the change of renal function during hospitalization. Gottlieb et al. have shown that even a small increase in serum creatinine, e.g., 0.1 mg/dl will worsen the outcome of the patients. It is also noteworthy that a significant rise in serum Cr generally may occur in the first 3 d of the admission to the hospital. The mortality rate in ADHERE registry is 4% for all the patients; however, the mortality of patients with significant renal insufficiency, i.e., Cr >3 mg/dl, is 9.4%, and the length of hospital stay is also lengthened as compared with those who do not have renal insufficiency. In another study of 1681 patients admitted for ADHF, Krumholz et al. found worsening renal function during hospitalization in 28% of patients. In-hospital mortality was more than double in those with versus without worsening renal function (7% versus 3%). This significant difference remained at 30 d (10% versus 6%) and 6 mo (25% versus 19%). The CHARM investigators also studied predictors of outcome in all three component trials in 2680 patients for an average of 34 mo. They found that every 10 ml/min decrease in eGFR increased the adjusted HR of cardiovascular death or readmission to the hospital by 10% (1.10, CI 1.07 to 1.13, P < 0.001). Therefore, even small changes in Cr have an important impact on in-patient mortality as well as postdischarge mortality.

Patients hospitalized for HF are at high risk for all-cause rehospitalization, with a 1-month readmission rate of 25% [4]. In 2013, physician office visits for HF cost $1.8 billion. The total cost of HF care in the United States exceeds $30 billion annually, with over half of these costs spent on hospitalizations [3]. Presently, HF is the leading cause of hospitalization among patients >65 years of age; the largest percentage of expenditures related to HF are directly attributable to hospital costs. Moreover, in addition to costs, hospitalization for acutely decompensated HF represents a sentinel prognostic event in the course of many patients with HF, with a high risk for recurrent hospitalization (50% at 6 months). Median length of in-hospital stay in the United States is approximately 4 days, whereas lengths of stay in Europe are generally markedly longer with a median of 9 days as reported in the EuroHeart Failure Survey II. Although systemic and pulmonary congestion is the main reason for hospitalization in most patients, many do not have a decrease in body weight during their hospital stay and are discharged with signs and symptoms of HF. Given that re-hospitalization drives much of the cost associated with HF, there has been increased interest in predicting risk of re-hospitalization as a means to control health care costs and reduce future risk. These risk stratification models can serve as important clinical tools by helping to identify those patients at both ends of the spectrum of risk; patients who are at very high risk may be observed more closely or treated more intensively, whereas patients at low risk may need less rigorous follow-up and monitoring. In the cohort from the OPTIMIZE-HF study with 60- to 90-day follow-up data, the most important predictors for the combined endpoint of death or re-hospitalization were admission serum creatinine concentration, systolic blood pressure, admission hemoglobin level, discharge use of ACE inhibitor or ARB, and pulmonary disease. In the EVEREST trial, composed of patients admitted with worsening HF and reduced ejection fraction, independent predictors during hospitalization of readmission and mortality included low admission Kansas City Cardiomyopathy Questionnaire score, high BNP, hyponatremia, tachycardia, hypotension, absence of beta blocker therapy, and history of diabetes and arrhythmias. Nevertheless, both models fail to provide the treating physician a simple decision making tool for predicting which patient is stable enough to be discharged from the hospital without a high risk of readmission. On this regard, high levels of BNP were found to be a reliable prognostic marker for HF patients readmission after discharge. Hospitalized patients with HF can be classified into important subgroups. These include patients with acute coronary ischemia, accelerated hypertension and acutely decompensated HF, shock, and acutely worsening right HF. Each of these various categories of HF has specific etiologic factors leading to decompensation, presentation, management, and outcomes. Noninvasive modalities can be used to classify the patient with hospitalized HF. The history and physical examination allows estimation of a patient's hemodynamic status, that is, the degree of congestion ("dry" versus "wet"), as well as the adequacy of their peripheral perfusion ("warm" versus "cold"). There have been limited previous randomized trials of therapy tailored during continuous hemodynamic monitoring in heart failure. Use of an indwelling pulmonary artery catheters to adjust therapy in advanced heart failure was first described by Kovick et al and subsequently by Pierpont for vasodilator therapy in decompensated heart failure with high systemic vascular resistance. There have been 11 additional randomized trials of PACs in critical care. A meta-analysis of these trials, including ESCAPE, showed that PAC was neutral in its effect on mortality and rehospitalization. These trials support the safety of PACs and the overall neutral effect, while highlighting the challenge of assessing a diagnostic tool without a consistent strategy of response with effective therapies. These results might be explained by the balance effect of improved treatment by tailored medicine that was counteracted by the invasive nature of PAC.

The Non-Invasive Cardiac System (NICaS: NI Medical, Hod-Hasharon, Israel), calculates the cardiac output (CO) by measuring whole body bio impedance in a tetra-polar mode, derived from electrodes placed on both wrists or one wrist and the contra-lateral ankle. This simple to operate, non-invasive technique was validated in several studies to be reliable in estimation of CO compared to traditional, invasive techniques in different settings including HF patients. A previous study demonstrated that parameters derived from this system showed a highly significant correlation to echocardiogram estimated ejection fraction and serum BNP in chronic HF patients and were equally able to predict complications in this population

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. HF admitted patient from cardiology and internal medicine departments in our institution.
3. Reduced EF ≤ 40%.
4. Elevated filling pressures, indicated by one symptom AND one physical sign: Symptoms : Dyspnea at rest, in the supine position, OR immediately upon routine activity, abdominal discomfort, severe anorexia, or nausea without apparent cause other than hepatosplanchnic congestion Signs: Jugular venous pressure elevation >10 cm above the right atrium, hepatomegaly, ascites, or edema in the absence of other obvious causes, rales greater than 1/3 lung fields, oxygen saturation < 90 % in room air, pulmonary venous congestion determined from chest x-ray films

Exclusion Criteria:

1. Severe aortic valve regurgitation and/or aortic stenosis.
2. Aortic aneurysm.
3. Heart rate above 130 beats/min.
4. Intra- and extra-cardiac shunts.
5. Severe peripheral vascular disease.
6. Severe pitting edema.
7. Sepsis.
8. Use of hemodialysis.
9. Patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Renal function deterioration during hospitalization | 6 months
  Renal function deterioration during hospitalization - worsening renal function (defined as an increase in the serum creatinine level of more than 0.3 mg per deciliter) at any time from randomization to dischage.

SECONDARY OUTCOMES:
30 days rehospitalization due to decompensated heart failure | 30 days
  30 days rehospitalization due to decompensated heart failure
Length of hospitalization | 3 months
  Length of hospitalization
All cause mortality at 30 days | 30 days
  All cause mortality at 30 days
All cause mortality at 3 months | 3 months
  All cause mortality at 3 months
All cause rehospitalization at 3 months | 3 months
  All cause rehospitalization at 3 months
Heart failure rehospitalization at 3 months | 3 months
  Heart failure rehospitalization at 3 months
Weight Loss during hospitalization - changes in body weight and net fluid loss | 5 days
  Weight Loss during hospitalization - changes in body weight and net fluid loss
Health-Related Quality of Life and Functional Status - patient-reported dyspnea | 3 months
  Health-Related Quality of Life and Functional Status - patient-reported dyspnea
Usage of mechanical ventilation | 5 days
  Usage of mechanical ventilation
Change in BNP/ pro-BNP from baseline to discharge Peak Troponin during the hospitalization | 5 days
  Change in BNP/ pro-BNP from baseline to discharge Peak Troponin during the hospitalization
Free from congestion (defined as jugular venous pressure of <8 cm, with no orthopnea and with trace peripheral edema or no edema) at 72 hours | 72 hours
  Free from congestion (defined as jugular venous pressure of <8 cm, with no orthopnea and with trace peripheral edema or no edema) at 72 hours
Emergency room visit within 60 days | 60 days
  Emergency room visit within 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Arbel, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel